CLINICAL TRIAL: NCT06585553
Title: Patients with Intestinal Metaplasia in the Lesser Curvature of the Gastric Corpus Require OLGIM Staging: a Secondary Analysis of a Prospective Cohort
Brief Title: Atrophic Gastritis and OLGIM Stage
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, professor, Shandong University
Other Study IDs: 20240904
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Intestinal Metaplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- atrophic gastritis: Perform Kimura-Takemoto and OLGIM staging

SUMMARY:
Three clinical research coordinators recruited patients aged 40-75 who underwent screening endoscopy at the Digestive Endoscopy Center of Qilu Hospital from July 1, 2022, to July 30, 2024. All participating patients provided written informed consent. Baseline information such as height, weight, age, sex, smoking and alcohol consumption status, HP status, and family history of gastrointestinal tumors were recorded before endoscopy. During endoscopy, the endoscopist observed and photographed the lesser and greater curvature of the antrum, corpus, and incisura, performed the Kimura-Takemoto classification, and classified those with a Kimura-Takemoto score of C0 as non-atrophic gastritis and those with C1-O3 as atrophic gastritis. Patients with atrophic gastritis received free multiple-site biopsies for pathological assessment, including targeted biopsies of suspected IM areas and random biopsies from Sydney classification sites. At least four biopsies were taken from the lesser and greater curvature of the antrum and corpus for pathological evaluation, and OLGIM staging was calculated based on the results.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were patients aged 40-75 undergoing painless screening endoscopy

Exclusion Criteria:

1) previous gastric surgery; 2) inability to undergo biopsy due to anticoagulant use; 3) refusal to sign informed consent; 4) history of radiotherapy or chemotherapy; 5) new diagnosis of advanced gastric cancer during endoscopy; 6) failure to complete multiple-site biopsy for atrophic gastritis; and 7) diagnosis of non-atrophic gastritis during endoscopy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the gastrointestinal endoscopy examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 2121 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic Performance of IM at Different Sites | 3 years
  Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of IM at different gastric sites for predicting OLGIM stage III/IV were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Jinan, Shandong, China